CLINICAL TRIAL: NCT06357702
Title: Initial Evidence for a Brief Psychological Telehealth Intervention for Patients With Chronic Masticatory Muscle Pain
Brief Title: K23- Physical Self Regulation vs Placebo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ian Boggero, PhD (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor-Investigator, Ian Boggero, PhD, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81313; K23DE031807 (NIH)
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Disorder
Keywords: myalgia; orofacial; telehealth
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Self Regulation (Experimental): 2 experimental telehealth sessions approximately 2 weeks apart
  Interventions: Behavioral: Physical Self Regulation Telehealth
- Psycho-education (Active Comparator): 2 control telehealth sessions approximately 2 weeks apart
  Interventions: Behavioral: Psycho-education Telehealth

INTERVENTIONS:
Behavioral: Physical Self Regulation Telehealth — 2 sessions of an intervention delivered via telehealth. Session 1 includes awareness and strategies for monitoring habits and 4 exercises to practice 5 times per day. Session 2 will be 2 weeks later and is a review of session 1 and an introduction to diaphragmatic breathing. Breathing is practiced for 15 minutes twice per day.
  Other Names: PSR-TH
  Arms: Physical Self Regulation
Behavioral: Psycho-education Telehealth — 2 sessions of an intervention delivered via telehealth. Session 1 includes discussing trigeminal nerve function, jaw and muscle anatomy, posture, pain referral patterns, and stress biology. Participants rate pain and jaw fatigue 5 times per day. Session 2 will be 2 weeks later and consists of checking on the homework and information from session 1,followed by a discussion of autonomic nervous system activity, and a discussion of sleep quality and sleep hygiene. Participants will be instructed to rate their stress levels, pain, and mood several times per day, similar to the times when participants in the PSR-TH condition would be practicing diaphragmatic breathing
  Other Names: Control
  Arms: Psycho-education

SUMMARY:
This study will use a between-person design. Participants will be treatment-seeking patients with chronic masticatory muscle pain. Participants who are eligible for the study and consent to participate will be randomly assigned to receive a brief behavioral intervention for chronic orofacial pain called Physical Self-Regulation or a control intervention. Interventions will be administered via telehealth in both arms. Both interventions will consist of 2 50-minute sessions scheduled approximately two weeks apart. Participants will be contacted two weeks and three months after completing the interventions to provide additional follow-up data. Investigators hypothesize that both PSR-TH and the control intervention will demonstrate strong feasibility (i.e., recruitment of at least 1 participant per week, >75% retention, >95% interventionist fidelity, and adequate acceptability, credibility, and burden). Investigators also hypothesize that specific biopsychosocial variables will moderate PSR-TH-related changes in outcomes, and that PSR-TH-related changes in perceived control over pain, self-efficacy, coping, parafunctional habits, and relaxation will mediate treatment effects.

DETAILED DESCRIPTION:
Chronic masticatory muscle pain disorders (MMPD) consist of several conditions (e.g., myofascial pain, local myalgia) characterized by pain in the muscles of the temporomandibular area lasting longer than three months. MMPD affects 5-12% of adults, is the most common cause of chronic non-odontogenic facial pain, and the second most common musculoskeletal pain condition after chronic low back pain. MMPD is associated with pain-related interference with daily activities, diminished quality of life (QoL) and costs of > $4 billion/year in the US, representing a serious public health issue. Chronic MMPD is most effectively managed with multidisciplinary treatment. One brief psychological intervention that has been particularly promising for improving orofacial pain outcomes and QoL in MMPD is physical self-regulation (PSR). Relative to standard dental care (SDC) alone, those who received SDC+PSR experienced reduced pain intensity up to 6.5 months later (Cohen's D = 0.67). These data suggest that PSR may be a promising intervention for improving pain outcomes in MMPD. Despite the promise of PSR, one of its major shortcomings is that treatment utilization is low, with less than 50% of eligible patients beginning PSR when offered in person. Offering PSR via telehealth may be a solution. Telehealth interventions improve access to care and are preferred by patients over in-person interventions. Preliminary data of treatment utilization for PSR-TH are promising, with over 80% of eligible patients beginning the intervention when offered via telehealth. However, it is not known if PSR-TH is efficacious above and beyond nonspecific treatment effects (e.g., people having more contact with a therapist, people inadvertently modifying their behavior to please their therapist, natural regression to the mean of pain symptoms, etc.). The efficacy of PSR-TH to treat MMPD needs to be formally tested; however, additional data regarding feasibility and moderating/mediating factors of PSRTH are needed to support such a trial. First, PSR-TH and a control intervention need to be formally piloted in patients with MMPD to 1) determine how willing patients are to participate in research (i.e., recruitment), 2) determine the completion rates for both interventions (i.e., retention), 3) quantify how well interventionists are able to deliver the interventions in a standardized way (i.e., fidelity), and 4) establish patients' perceived acceptability, credibility, and burden of both interventions. Second, a body of work has examined biopsychosocial moderators and mediators of responses to psychological interventions (e.g., cognitive behavioral therapy, [CBT]) in MMPD, but never of PSR-TH specifically. Identifying relevant moderators and mediators in this project will allow for more thorough assessment of those specific relationships in a future Phase II trial, advancing understanding of how PSR-TH works, and for whom. To accomplish these aims, treatment-seeking patients with chronic MMPD will be randomly assigned to two 50-min telehealth sessions of PSR or a control intervention (N=52/group) and will provide biopsychosocial moderator, mediator, and outcome data at baseline, after each intervention sessions, two weeks following the intervention, and three months following the intervention. The investigators hypothesize that both PSR-TH and the control intervention will demonstrate strong feasibility (i.e., recruitment of at least 1 participant per week, >75% retention, >95% interventionist fidelity, and adequate acceptability, credibility, and burden). The investigators also hypothesize that specific biopsychosocial variables will moderate PSR-TH-related changes in outcomes, and that PSR-TH-related changes in perceived control over pain, self-efficacy, coping, parafunctional habits, and relaxation will mediate treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary or secondary chronic masticatory muscle pain diagnosis
* Provide signed and dated electronic informed consent form
* Willing to comply with all study procedures
* Male or female, aged 18 or over
* Be able to speak and write in English
* Be seeking treatment at UKOPC
* Have the ability to perform telehealth visits (i.e., internet access, phone, tablet, computer or other device with audio/visual capabilities)

Exclusion Criteria:

* Currently using anticonvulsant, steroid, antispasmodic, or opioid medication for chronic pain 2 days a week or more often
* Have current or recent (within the last 3 months) psychotic, suicidal, homicidal, or manic symptoms. Participants with a history of such symptoms must demonstrate psychiatric stability for at least 6 months and be under the care of a medical or mental health professional for symptom management prior to being eligible for the study (must have written note from physician authorizing them to participate)
* Patients who are currently on medication for diabetes or seizures (i.e., epilepsy) must have written clearance from their medical providers prior to participating in the study
* History of seizures within the last 12 months
* Pain duration less than 3 months
* Pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline (week 0), post intervention (week 5) and 3-month follow-up (week 15)
  Pain intensity will be measured with the Graded Chronic Pain Scale Pain Intensity Subscale. Participants rate their worst pain, least pain, average pain, in the last 24 hours and pain right now using an 11 point Likert scale ranging from 0 to 10 with higher scores equating to greater pain. Scores are averaged for the total pain intensity score.
Change in pain interference | Baseline (week 0), post intervention (week 5) and 3-month follow-up (week 15)
  Pain interference will be measured with the The Graded Chronic Pain Scale Pain Interference Subscale. Participants rate how much the pain has interfered with 7 daily activities on an 11 point Likert scale ranging from 0 to 10 with higher scores equating to greater interference. Pain interference is scored as the mean of the 7 items.
Change in quality of life | Baseline (week 0), post intervention (week 5) and 3-month follow-up (week 15)
  Quality of life will be measured with the Satisfaction with Life Scale. Likert scale with 7 items scores range from 7 to 35 with higher scores equating to better quality of life.
Recruitment rate | Baseline (week 0)
  Number of patients who are consented into the study per month
Retention rate | Follow up Visit at Month 3 (week 15)
  Number of consented patients who also complete the three-month follow-up assessment
Interventionist Fidelity Session 1 | Study Visit 1 (week 1)
  Each intervention session will have a checklist of items that need to be covered by the interventionists. All study sessions will be audio-recorded. A subset of all audio recordings will be checked for interventionist fidelity, defined by the following percentage:
  Total items covered by interventionist/ Total possible items to be covered in that session
Interventionist Fidelity Session 2 | Study Visit 2 (week 3)
  Each intervention session will have a checklist of items that need to be covered by the interventionists. All study sessions will be audio-recorded. A subset of all audio recordings will be checked for interventionist fidelity, defined by the following percentage:
  Total items covered by interventionist/ Total possible items to be covered in that session
Treatment Acceptability | Study Visits 1 and 2 (up to 2 weeks)
  Treatment Acceptability and Adherence Scale. The scale will measure what participants overall evaluation of if treatment was fair, reasonable, and appropriate. 6 item Likert scale with scores on each item ranging from 1 to 9 with higher scores equating to greater acceptability. Acceptability is scored as the mean of the 6 items.
Treatment Credibility | Study Visits 1 and 2 (up to 2 weeks)
  Treatment Credibility/Expectancy Scale will measure how feasible is it the intervention will work and work for the participant.
  6 item Likert scale with scores on each item ranging from 1 to 9 with higher scores equating to greater credibility. Acceptability is scored as the mean of the 6 items.
Research Burden | Follow up Visit at Month 3 (week 15)
  Research burden will be measured by administering 8 selected items from the Perceived Research Burden Assessment. Participants rate how burdensome the study was on an 8 item assessment on a 5 point Likert scale ranging from strongly disagree to strongly agree with higher scores equating to greater burden. Burden is scored as mean of the 8 items.

SECONDARY OUTCOMES:
Treatment Satisfaction | 2-week follow-up (week 5)
  Treatment Satisfaction Questionnaire 8 items on a 4 point Likert scale. Higher scores equate to greater satisfaction. Satisfaction is scored as mean of the 8 items.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Boggero, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No